CLINICAL TRIAL: NCT03244254
Title: I-FABP Levels in Pediatric Celiac Patients in Transition From Active Disease to Remission
Brief Title: Intestinal Fatty Acid-binding Protein (I-FABP) Levels in Pediatric Celiac Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Schneider Children's Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr. Assaf Hoofien, Research fellow, Schneider Children's Medical Center, Israel
Other Study IDs: SchneiderCMCIsraelIFABP
Record Dates: First submitted 2017-08-06; First posted 2017-08-09 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Celiac Disease in Children
Keywords: Celiac Disease; Children; I-FABP
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test Group: Children up to 17 years of age at recruitment undergoing endoscopy in order to diagnose or rule out Celiac disease, whose Marsh score at endoscopy is 2 or higher.
- Control Group: Children up to 17 years of age undergoing endoscopy as part of abdominal pain workup, whose Celiac serology is negative, and the Marsh score found at endoscopy is 0.

SUMMARY:
A prospective, longitudinal study meant to compare blood levels of I-FABP in pediatric celiac patients during diagnosis to levels under gluten free diet, it's correlation with traditional serology testing and questionnaire regarding patient responsiveness to the gluten free diet, and in comparison to a control group.

DETAILED DESCRIPTION:
I-FABP is a reliable marker for intestinal damage and has been proved to respond more swiftly than traditional serology to enterocyte injury in celiac patients who do not a gluten free diet. In this study a pediatric population of celiac patients will be tested for I-FABP levels during initial endoscopic diagnosis and during one year of follow up. Their levels will be compared to a control group of pediatric patients undergoing endoscopy for reasons other than suspicion of celiac disease. During the period of follow up, the test group will undergo repeat testing for I-FABP levels, as well as the traditional follow up testing for serology in celiac patients and a questionnaire regarding. The results will be analyzed in the hope of finding a way to use I-FABP as a more direct, accurate marker of disease activity, and of correlations between it's level and the patient's Marsh score at diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing endoscopy for diagnosis of celiac disease, with elevated serology (TTG more than 3 times the norm), and whose histological Marsh score is 2 or higher.

Exclusion Criteria:

* Diseases known to cause elevation in I-FABP levels: Bowel ischemia, inflammatory bowel disease, Primary Biliary Cholangitis, liver failure, biliary duct obstruction, liver malignancy.
* Bowel trauma or abdominal surgery or acute gastroenteritis in the last 3 months
* NSAID use in the last week.
* Intensive daily physical activity (over 1 hour) in the 2 days prior to endoscopy.
* Known genetic disorders (such as Down's syndrome).
* Patients whose TTG was elevated but lower than 3 times the normal range.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients undergoing endoscopy at the research hospital.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
I-FABP levels at diagnosis | 1 day of enrollment
  Comparison of I-FABP levels at day of enrollment (and endoscopy) between test and control groups.
I-FABP levels during remission | 6 months & 12 months after enrollment
  Follow-up of I-FABP levels in test groups during follow-up meetings, comparison with other celiac serology taken at follow-up and adherence to gluten free diet (measured using adherence questionnaires)

CONTACTS AND LOCATIONS:
Overall Officials: Raanan Shamir, Prof, Study Director — Director
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel